CLINICAL TRIAL: NCT01396096
Title: Comparison of Obesity Alleles Among Diverse Demographic Patient Populations Undergoing Bariatric Surgery
Brief Title: Comparison of Obesity Alleles Among Diverse Demographic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00634
Record Dates: First submitted 2011-07-12; First posted 2011-07-18 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from 0.35ml of EDTA-anticoagulated whole blood using the Qiagen MagAttract DNA Blood Midi M48 Kit and Qiagen BioRobot M48 Workstation (Qiagen, Valencia, California) according to the manufacturer's directions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This proposal is designed to (1) establish the feasibility of a research strategy for discovering ethnic differences in the frequency of genotypes in patients after bariatric surgery and (2) perform a preliminary evaluation of this research strategy. Our goal is to identify genetic factors that may influence the success of various surgical weight loss interventions and determine whether these factors are associated with specific patient populations.

DETAILED DESCRIPTION:
Goals:

1. Establish feasibility of obtaining research consent on patients to collect clinical data, family history, and blood samples.
2. Complete comprehensive genetic analyses on a diverse group of severely obese patients who have undergone bariatric surgery, specifically the primarily non-Caucasian Bellevue population and the Caucasian population of Geisinger Health Systems and NYU Langone Weight Management Program, to help define genetic factors that influence which surgical interventions work best for which patients. The ultimate aim is to rapidly translate these discoveries into practical solutions.

Methods and Procedures: The participants of this study are all patients who have undergone bariatric surgery at Bellevue Hospital, NYU Langone Weight Management Program, and Geisinger Health System. The investigators have already completed this in 200 patients and plan to increase enrollment for a total of 2500 patients. The investigators will collect blood samples on bariatric surgery patients and send the blood to Geisinger for genotyping and analysis. An extra sample of venous blood (about 4 tablespoons or 40ml) will be collected at the time of routine postoperative visits. In addition, the investigators will use information that has routinely been and will be collected during postoperative visits as part of the care that bariatric patients receive. The investigators will look at the electronic medical record to obtain the preoperative weights. This includes questionnaires patients complete and the results of the laboratory tests and other studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone any type of bariatric surgery

Exclusion Criteria:

* Patients who have not had bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NYUMC/Bellevue: All patients seen in the Bariatric Surgery Program at Bellevue NYU Langone Weight Management Program: All patients who are at least post-op 2 years
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Complete comprehensive genetic analyses | 01/01/2016

CONTACTS AND LOCATIONS:
Overall Officials: Manish Parikh, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Background] Walley AJ, Blakemore AI, Froguel P. Genetics of obesity and the prediction of risk for health. Hum Mol Genet. 2006 Oct 15;15 Spec No 2:R124-30. doi: 10.1093/hmg/ddl215. PMID 16987875